CLINICAL TRIAL: NCT05112159
Title: A Phase 1, First-in-human, Randomized, Double-blind, Placebo-controlled, Single Dose Escalation Study to Evaluate the Safety, Tolerability, and Pharmacokinetics (PK) of Orally Administered IPG1094 in Healthy Adult Participants
Brief Title: Study of IPG1094 in Healthy Participants
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanjing Immunophage Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IPG1094-A001
Record Dates: First submitted 2021-09-16; First posted 2021-11-08 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-10

CONDITIONS: Safety Issues
Keywords: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- IPG1094 100mg (Experimental): Four subjects in this cohort will receive a single dose of IPG1094 100 mg qd and two subjects will receive a single dose of placebo 100mg qd orally. Sentinel subjects (i.e. 1 subject will be dosed with IPG1094 and 1 with placebo before the remainder of the cohort is dosed) will be used in the cohort.
  Interventions: Drug: IPG1094; Drug: placebo
- IPG1094 300mg (Experimental): Six subjects in this cohort will receive a single dose of IPG1094 300 mg qd and two subjects will receive a single dose of placebo 300mg qd orally.
  Interventions: Drug: IPG1094; Drug: placebo
- IPG1094 600mg (Experimental): Six subjects in this cohort will receive a single dose of IPG1094 600 mg qd and two subjects will receive a single dose of placebo 600mg qd orally.
  Interventions: Drug: IPG1094; Drug: placebo
- IPG1094 900mg (Experimental): Six subjects in this cohort will receive a single dose of IPG1094 900 mg qd and two subjects will receive a single dose of placebo 900mg qd orally.
  Interventions: Drug: IPG1094; Drug: placebo
- IPG1094 1200mg (Experimental): Six subjects in this cohort will receive a single dose of IPG1094 1200 mg qd and two subjects will receive a single dose of placebo 1200 mg qd orally.
  Interventions: Drug: IPG1094; Drug: placebo
- IPG1094 1500mg (Experimental): Six subjects in this cohort will receive a single dose of IPG1094 1500 mg qd and two subjects will receive a single dose of placebo 1500mg qd orally.
  Interventions: Drug: IPG1094; Drug: placebo

INTERVENTIONS:
Drug: IPG1094 — The IPG1094 drug product is supplied as oral tablet dosage form, containing two strengths: 50 mg and 100 mg, respectively, which contain IPG1094.
Drug: placebo — Matching placebo tablets to IPG1094 50mg and 100mg

SUMMARY:
This is a phase 1, first-in-human, randomized, double-blind, placebo-controlled, single dose escalation study to evaluate the safety, tolerability, and PK of single dose orally administered IPG1094 in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following criteria to be included in the study:

Demography

1. Healthy adult male or female participants between 18 and 50 years of age (inclusive).
2. Body weight between 50 and 100 kg (inclusive) and body mass index (BMI) within 18~32 kg/m2 (inclusive).

   Health status
3. In good health as determined by screening tests. Good health is defined as having no clinically relevant abnormalities identified by a detailed medical history, full physical examination (including measurement of blood pressure and pulse rate), 12-lead ECG, and clinical laboratory tests.

   Vital signs (measured after resting for 5 minutes seated position) within normal range, or outside the normal range and not considered clinically significant by the Investigator.

   Standard 12-lead ECG parameters (recorded after resting for 5 minutes in supine position) in the following ranges; corrected QT interval(QTc) (Fridericia algorithm recommended) ≤ 450 ms for males and 470 ms for females, and normal ECG tracing, or abnormal ECG tracing not considered clinically relevant by the Investigator.

   Laboratory parameters demonstrating no clinically significant abnormalities, as determined by the Investigator. A total bilirubin outside the normal range may be acceptable if total bilirubin does not exceed 1.5 × upper limit of normal(ULN) conjugated bilirubin (with the exception of a participant with documented Gilbert syndrome).
4. A negative result on urine drug screen and a repeat negative result on Day -1 (amphetamines/methamphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, opiates).
5. Female participants must not be pregnant or breastfeeding and must use an effective contraception method (as described in Section 4.5.4), with the exception of participants who have undergone sterilization in the preceding 3 months, or who are postmenopausal.

   A woman of childbearing potential (WOCBP) must undergo pregnancy testing prior to the first dose of the Investigational Medicinal Product (IMP). The participant must be excluded from the study if the serum pregnancy test is positive.

   A postmenopausal state is defined as 12 months of amenorrhea without an alternative medical cause. In the absence of 12 months of amenorrhea, menopause may be confirmed by follicle stimulating hormone（FSH） measurement (> 40 IU/L or milli-International unit（mIU）/mL).Females on Hormonal Replacement therapy (HRT ), where menopausal status is indeterminate, will be required to use a non-estrogen hormonal contraceptive method if participants wish to continue their HRT during the study. Participants must otherwise discontinue HRT to allow for confirmation of postmenopausal status prior to enrollment in the study.

   Regulation
6. Provide written informed consent prior to undertaking any study-related procedures.
7. Must not be under any administrative or legal supervision or under institutionalization as per a regulatory or juridical order.

Exclusion Criteria:

Participants who meet any of the following criteria will be excluded from the study:

Medical history and clinical status

1. Any history or presence of clinically relevant cardiovascular, pulmonary, gastrointestinal, hepatic, renal, metabolic, hematological, neurological, musculoskeletal, rheumatological, psychiatric, systemic, ocular, or infectious disease, or signs of acute illness.
2. Frequent severe headaches and/or migraines, recurrent nausea and/or vomiting (defined as vomiting more than twice a month).
3. Made a blood donation of any volume within 2 months prior to the first dose.
4. Symptomatic postural hypotension, irrespective of actual decrease in blood pressure, or asymptomatic postural hypotension with a decrease in systolic blood pressure ≥30 mmHg within 3 minutes of moving from supine to standing position.
5. Presence or history of drug hypersensitivity, or anaphylactic reaction, diagnosed and treated by a physician.
6. Known hypersensitivity to any component of the IMP formulation.
7. History or presence of drug or alcohol abuse (defined as alcohol consumption more than 2 units per day on a regular basis).
8. Regular smoking (defined as more than 5 cigarettes or equivalent per week), or unable to stop smoking during the study. Occasional smokers may be enrolled.
9. Excessive consumption of beverages containing xanthine bases (defined as more than 4 glasses per day).

   Interfering substances
10. Any medication, including St John's Wort, within 14 days prior to administration of the first dose or within 5 times the elimination half-life or pharmacodynamic half-life of the medication, with the exception of hormonal contraception, menopausal hormone replacement therapy, or occasional paracetamol at doses up to 2g/day.
11. Any consumption of grapefruit or products containing grapefruit within 5 days prior to the first dose administration.
12. Any vaccination in the 28 days prior to administration of the first dose.

    General conditions
13. Any participant who, in the judgment of the Investigator, is likely to be non-compliant during the study, or to be unable to cooperate due to language problems or poor mental development.
14. Any participant who enrolled in or participated in any other clinical study involving an investigational medicinal product, or in any other type of medical research within 1 month or within 5 times the elimination half-life prior to administration of the first dose.
15. Any participant who cannot be contacted in the case of an emergency.
16. Any participant who is the Investigator or any sub-investigator, research assistant, pharmacist, study coordinator, or other staff thereof directly involved in conducting the study or any person dependent on (employees or immediate family members) the study site, the Investigator or the Sponsor.

    Biological status
17. Positive result on any of the following tests: hepatitis B surface antigen (HBsAg), hepatitis B core antibodies (HBcAb), anti-hepatitis C virus antibodies (anti-HCV), anti-human immunodeficiency virus 1 and 2 antibodies（anti-HIV1 and anti-HIV2 Ab).
18. Positive alcohol test.
19. Any participant in whom venous blood collection is difficult.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2021-09-27 (Actual); Primary Completion 2022-05-18 (Estimated); Study Completion 2022-07-30 (Estimated)

PRIMARY OUTCOMES:
Occurrence of all adverse events | Up to 8 days
  Evaluation of adverse events
RBC | Up to 8 days
  Evaluation of Hematology
white blood cell count (WBC) | Up to 8 days
  Evaluation of Hematology
platelet count (PLT) | Up to 8 days
  Evaluation of Hematology
haemoglobin (HGB) | Up to 8 days
  Evaluation of Hematology
mean corpuscular hemoglobin | Up to 8 days
  Evaluation of Hematology
mean corpuscular hemoglobin concentration | Up to 8 days
  Evaluation of Hematology
Hematocrit | Up to 8 days
  Evaluation of Hematology
mean corpuscular volume (MCV) | Up to 8 days
  Evaluation of Hematology
absolute differential leukocyte count (eosinophils) | Up to 8 days
  Evaluation of Hematology
absolute differential leukocyte count (monocytes) | Up to 8 days
  Evaluation of Hematology
absolute differential leukocyte count (lymphocytes) | Up to 8 days
  Evaluation of Hematology
absolute differential leukocyte count (basophils) | Up to 8 days
  Evaluation of Hematology
absolute differential leukocyte count (neutrophils) | Up to 8 days
  Evaluation of Hematology
Temperature (°C ) | Up to 8 days
  Evaluation of Vital Signs
Respiration rate | Up to 8 days
  Evaluation of Vital Signs
Pulse rate | Up to 8 days
  Evaluation of Vital Signs
Blood pressure (both systolic and diastolic) | Up to 8 days
  Evaluation of Vital Signs
Standard 12-lead ECG - heart rate | Up to 8 days
  Evaluation of Electrocardiograms
Standard 12-lead ECG - QTcF | Up to 8 days
  Evaluation of Electrocardiograms
Standard 12-lead ECG - PR | Up to 8 days
  Evaluation of Electrocardiograms
Standard 12-lead ECG - QRS | Up to 8 days
  Evaluation of Electrocardiograms
Standard 12-lead ECG - QT | Up to 8 days
  Evaluation of Electrocardiograms
Alanine aminotransferase (ALT) | Up to 8 days
  Evaluation of Serum Chemistry
albumin (ALB) | Up to 8 days
  Evaluation of Serum Chemistry
alkaline phosphatase (ALP) | Up to 8 days
  Evaluation of Serum Chemistry
aspartate aminotransferase (AST) | Up to 8 days
  Evaluation of Serum Chemistry
total bilirubin (TBil) | Up to 8 days
  Evaluation of Serum Chemistry
Urea | Up to 8 days
  Evaluation of Serum Chemistry
calcium (Ca) | Up to 8 days
  Evaluation of Serum Chemistry
chloride (Cl) | Up to 8 days
  Evaluation of Serum Chemistry
cholesterol (CHO) | Up to 8 days
  Evaluation of Serum Chemistry
creatinine (Cr) | Up to 8 days
  Evaluation of Serum Chemistry
creatine kinase (CK) | Up to 8 days
  Evaluation of Serum Chemistry
glucose (Glu) | Up to 8 days
  Evaluation of Serum Chemistry
lactate dehydrogenase (LDH) | Up to 8 days
  Evaluation of Serum Chemistry
phosphate (P) | Up to 8 days
  Evaluation of Serum Chemistry
potassium (K) | Up to 8 days
  Evaluation of Serum Chemistry
sodium (Na) | Up to 8 days
  Evaluation of Serum Chemistry
total protein (TP) | Up to 8 days
  Evaluation of Serum Chemistry
Prothrombin time (PT) | Up to 8 days
  Evaluation of Serum Coagulation
activated partial thromboplastin time (APTT) | Up to 8 days
  Evaluation of Serum Coagulation
fibrinogen | Up to 8 days
  Evaluation of Serum Coagulation
international normalized ratio (INR) | Up to 8 days
  Evaluation of Serum Coagulation
pH | Up to 8 days
  Evaluation of Urinalysis
Bilirubin (U-BIL) | Up to 8 days
  Evaluation of Urinalysis
glucose (GLU) | Up to 8 days
  Evaluation of Urinalysis
urine erythrocytes (U-RBC) | Up to 8 days
  Evaluation of Urinalysis
ketones (U-KET) | Up to 8 days
  Evaluation of Urinalysis
Urinary leukocyte (U-LEU) | Up to 8 days
  Evaluation of Urinalysis
nitrites (U-NIT) | Up to 8 days
  Evaluation of Urinalysis
protein (U-PRO) | Up to 8 days
  Evaluation of Urinalysis
specific gravity (U-SG) | Up to 8 days
  Evaluation of Urinalysis
urobilinogen (URO) | Up to 8 days
  Evaluation of Urinalysis

SECONDARY OUTCOMES:
Maximum plasma concentration（Cmax） | Blood samples will be collected at 0 h before administration (within 1h prior to administration), 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 9, 12, 24, 36, 48, 72, and 96 h after administration.
  Pharmacokinetic (PK) parameters after a single oral dose of IPG1094
Time to Cmax (tmax) | Blood samples will be collected at 0 h before administration (within 1h prior to administration), 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 9, 12, 24, 36, 48, 72, and 96 h after administration.
  Pharmacokinetic (PK) parameters after a single oral dose of IPG1094
Area under the serum concentration-time curve (AUC[0-t] | Blood samples will be collected at 0 h before administration (within 1h prior to administration), 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 9, 12, 24, 36, 48, 72, and 96 h after administration.
  Pharmacokinetic (PK) parameters after a single oral dose of IPG1094
Area under the serum concentration-infinity curve AUC[0-infinity] | Blood samples will be collected at 0 h before administration (within 1h prior to administration), 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 9, 12, 24, 36, 48, 72, and 96 h after administration.
  Pharmacokinetic (PK) parameters after a single oral dose of IPG1094
Apparent terminal phase half-life (t1/2) | Blood samples will be collected at 0 h before administration (within 1h prior to administration), 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 9, 12, 24, 36, 48, 72, and 96 h after administration.
  Pharmacokinetic (PK) parameters after a single oral dose of IPG1094

CONTACTS AND LOCATIONS:
Overall Officials: Wang Jianfei, Study Director — Nanjing Immunophage Biotech Co., Ltd
Locations (1):
- Scientia Clinical Research Ltd, Randwick, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No